CLINICAL TRIAL: NCT06391983
Title: Effect of Resistance Training on Intermuscular Adipose Tissue in Patients With Type 2 Diabetes
Brief Title: The Impact of Moderate Resistance Training on IMAT in Elderly Diabetes Patients Without Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lou Qingqing (Other Government)
Responsible Party: Sponsor-Investigator, Lou Qingqing, M.D. Director，Hainan Clinical Medical Research Center for Metabolic Disease, The First Affiliated Hospital of Hainan Medical University
Organization: The First Affiliated Hospital of Hainan Medical University (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LouQingqing
Record Dates: First submitted 2023-12-29; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- resistance training (Experimental): The intervention group attended online group education sessions on diabetes self management, as well as resistance exercise training sessions three times weekly; the sessions were approximately 40 minutes long and included 5 minutes of warm up, followed by 30 minutes of resistance exercises and 5 minutes of cool down. The resistance training consisted of ten upper-body and lower-body exercises using elastic band. The initial sessions were 1 to 2 sets of 6 to 8 repetitions at 45% of the one-repetition maximum (1 RM). It was increased progressively to 2 to 3 sets of 8 to 12 repetitions at approximately 55% of 1 RM. The 10 resistance exercises were reported elsewhere. Due to the Covid-19 pandemic, the participants performed resistance exercise at home, and 10 specific teaching videos (one video for each exercise) were provided for participants in this group. Wechat was used for attendance taking and communication.
  Interventions: Other: resistance training (elastic band)
- Control Group (Experimental): The control group was not asked to participate in any regular exercise. However, the group attended online group educational sessions about diabetes self management once a month, and were asked to record their daily physical activities. Online mini program Wechat was used for communication.
  Interventions: Other: resistance training (elastic band)

INTERVENTIONS:
Other: resistance training (elastic band) — The intervention group attended online group education sessions on diabetes self management, as well as resistance exercise training sessions three times weekly; the sessions were approximately 40 minutes long and included 5 minutes of warm up, followed by 30 minutes of resistance exercises and 5 minutes of cool down. The resistance training consisted of ten upper-body and lower-body exercises using elastic band. The initial sessions were 1 to 2 sets of 6 to 8 repetitions at 45% of the one-repetition maximum (1 RM). It was increased progressively to 2 to 3 sets of 8 to 12 approximately 50% -55% of 1 RM.

SUMMARY:
Data shows that high intensity resistance training reduces Intermuscular Adipose Tissue (IMAT) in obesity adults. Whether moderate resistance training reduces IMAT for non-obese elderly patients with diabetes is not clear. Therefore, this study aimed to evaluate the impact of moderate resistance training on IMAT in elderly patients with type 2 diabetes, and the independent effect of IMAT reduction on metabolic outcomes.

In this randomized control trial (RCT), 85 type 2 diabetes patients were randomized into the resistance training group (42 participants) and control group (43 participants) for 6-month intervention. The control group was not asked to participate in any regular exercise. However, the group attended online group educational sessions about diabetes self management once a month, and were asked to record their daily physical activities. Online mini program Wechat was used for communication. The intervention group attended online group education sessions on diabetes self management as the control group, as well as resistance exercise training sessions three times weekly; the sessions were approximately 40 minutes long and included 5 minutes of warm up, followed by 30 minutes of resistance exercises and 5 minutes of cool down. The resistance training consisted of ten upper-body and lower-body exercises using elastic band. The initial sessions were 1 to 2 sets of 6 to 8 repetitions at 45% of the one-repetition maximum (1 RM). It was increased progressively to 2 to 3 sets of 8 to 12 repetitions at approximately 50% -55% of 1 RM. The primary outcome were the changes of IMAT measured by computed tomography（CT）scan and magnetic resonance imaging (MRI) interactive decomposition of water and fat with echo asymmetry and least squares qualification sequence (IDEAL-IQ). The secondary outcomes were the changes in metabolic parameters.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* ≥60 and <75 years of age
* Normal muscle strength
* Body-mass index (BMI) ≤35
* Glycosylated hemoglobin A1c (HbA1c) < 9%

Exclusion Criteria:

* Patients who had severe chronic diabetes complications（e.g., stroke, myocardial infarction, end stage renal disease, proliferative retinopathy)
* Cognitive impairments

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
The primary outcome were the changes of IMAT | 6 months
  MRI IDEAL-IQ was used to quantitatively assess IMAT in the middle of left thigh.
  This study used fat fraction as the indicator to quantify IMAT of the thigh muscle.
  CT scan was used to assess IMAT area. Hounsfeild (Hu) was used to quantify the density of muscle or fat. The density of IMAT area is low, between -190Hu to -30Hu. With regard to muscle area, there are two different density areas: Normal attenuation muscle area, with density between 31Hu to 100Hu, representing normal muscle area, and Low attenuation muscle area, with density between 0Hu to 30Hu, representing fat infiltration, the lower the Hu, the higher the fat infiltration.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Hainan Medical University, Haikou, Hainan, China

IPD SHARING:
Plan to Share IPD: No